CLINICAL TRIAL: NCT00447252
Title: Needs Assessment for Bereaved Families
Acronym: NABF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herzog Hospital (Other)
Collaborators: Joint Distribution Committee (JDC) (Unknown)
Other Study IDs: Brom2CTIL
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Bereaved Families
Keywords: bereavement; grief

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The present study will focus on several objectives in the framework of the family perspective and systemic understanding of the mourning process:

1. Identification of the psychological, social and practical needs of families that have lost a child to terrorism.
2. Deepening and extending the knowledge of how families cope with the loss of a child in a violent incident of a security-related nature.
3. Identification of risk and resilience factors within the family structure, and the nature of the relationships within the family.

DETAILED DESCRIPTION:
Assessment of Families Who Have Undergone the Traumatic Loss of a Child Study Protocol

The present study will focus on several objectives in the framework of the family perspective and systemic understanding of the mourning process:

1. Identification of the psychological, social and practical needs of families that have lost a child to terrorism.
2. Deepening and extending the knowledge of how families cope with the loss of a child in a violent incident of a security-related nature.
3. Identification of risk and resilience factors within the family structure, and the nature of the relationships within the family.

The University of Al-Quds in East Jerusalem will be conducting an identical study in conjunction with this one, examining Palestinian families who have lost a child in the conflict with Israel. Collaboration between these studies will allow a cross-cultural comparison of family coping with traumatic loss, and of the identification of resilience and risk factors among the families.

Method of the study Participants. The assessment process will include some twenty-five Israeli families who have lost a son or daughter below the age of 18 as a result of a terrorist incident, at least six months previously. All family members living at home will participate in the study. The study will not include single-parent families, or family members who suffer from mental retardation, disturbances because of addiction, or psychiatric disturbance from the psychotic or autistic spectra (schizophrenia, manic-depressive illness, psychotic disturbances, PDD).

Procedure. The recruitment of families will be done by the Kobi Mandel Foundation, which is involved in helping families that have been victims of terror. The Foundation will not approach families who fit the criteria of ineligibility for the study, as described in the previous paragraph. The parents will fill out a form of informed consent on their own behalf, and on behalf of their children who are under the age of 18, after they have received an explanation about the procedure of the study, and have been given an opportunity to ask questions about it. Teenagers over 14 years old will sign a form of informed consent, with parental permission. Family members over the age of 18, living at home, will fill out a form of informed consent on their own behalf.

To carry out this stage, each family will be assigned a professional by the Israel Center for the Treatment of Psychotrauma, who will be its liaison and responsible for the process of assessment. The completion of the questionnaires will be coordinated with the family members, and carried out in the presence of the liaison, who will assist in explaining the questionnaire, and provide support in the event of emotional difficulties arising.

Every member of the family will fill out the questionnaire separately; the liaison will focus on helping children who have difficulty doing so. The parents will fill out questionnaires for small children (under 10 years old). In order to preserve the privacy of the participants, each family member will receive a personal code to be written on the questionnaire. The liaison alone will have the key to identify each participant, which is important for the identification of needs within the family, and the ability to direct them for appropriate treatment.

Possible risks. The main risk for the participants relates to the possible uncomfortable feeling the questionnaire might raise by evoking memories of the deceased, and to personal distress. For this reason, the questionnaires will be given to the participants by a trained professional who will be able to provide support, identify distress and suggest seeking professional treatment if necessary.

Qualifications of the Principal Investigators. The work will be carried out under the supervision of Dr. Danny Brom, the founder and current director of the Israel Center for the Treatment of Psychotrauma.

Description of the research instruments Demographic and organizational details. The participants will relate to demographic details like age, sex, family status, place in the family, occupation and socio-economic status, as well as information about the death (circumstances and time of death, description of the loss).

McMaster Family Assessment Device (FAD): This questionnaire contains 60 self-reported items that assess six aspects of family functioning: Problem solving, Communication, Roles, Affective responsiveness, Affective involvement, Behavior control In addition, the questionnaire contains a component (12 items) of general functioning (Epstein, Baldwin and Bishop, 1983).

Couple adjustment: Dyadic Adjustment Scale (DAS) (Spanier, 1976). The quality of mutual adjustment in the marital system will be measured by the DAS questionnaire, which contains 32 items in four subscales: Dyadic Consensus, Dyadic Satisfaction, Dyadic Cohesiveness and Affectional Expression.

Adults Grief Response: Inventory of Complicated Grief - ICG (Prigerson and Jacobs, 2001). The questionnaire examines adjustment to grief. Its 33 items measure non-adaptive symptoms of response to loss. The items make up two primary distress scales - traumatic distress and separation distress - which represent a uni-dimensional construct. The participants are asked to grade the degree to which they experience each of the symptoms presented, on a Likert scale of 1 (never) to 5 (always).

Exposure to trauma and post-traumatic distress. The PDS questionnaire (Foa, Feske & Murdock, 1993) will examine the history of traumatic events, subjective trauma response, post-traumatic symptoms and functional impairment. The questionnaire includes yes/no questions for the parent to answer regarding possible traumas in his or her past. Four yes/no questions examine the subjective response to the event (criterion A2). The section that examines post-traumatic symptoms includes 17 items that relate to the appearance of different symptoms, according to DSM, within the last month: re-experiencing the event (criterion B), avoidance (C) and hyperarousal (D). The scale of responses runs from 0 (not relevant or happened only once) to 3 (almost all the time). A grade of 2 or more is regarded as verifying the existence of a symptom.

Beyond this, the questionnaire contains nine yes/no questions that relate to impaired functioning in different areas of life, like work, relations with family members, leisure time activity, and so on.

Depression: Beck Depression Inventory (BDI-II). This widely accepted questionnaire measures the severity of symptoms of depression. It was updated in 1996 in order to meet the criteria of the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition). The participants are asked to relate to 21 items that describe different depressive symptoms on a scale of 0-3. A general score on the questionnaire can therefore lie between 0 and 63 (a higher score indicates greater severity of depressive symptoms).

Adolescents Grief response: UCLA Trauma Psychiatry Service Grief Inventory (Layne et al, 1998). On this questionnaire, the participants are required to answer ten items that relate to loss response, from 0 (not at all) to 4 (very much) on a Likert scale.

Post-traumatic symptoms. UCLA PTSD Reaction Index Adolescent Version (RI-R) (Rodriguez, Steinberg, & Pynoos, 1999). The RI-R is a new version of the earlier UCLA Reaction Index (Frederick, Pynoos, & Nader,1992), which was based on the DSM-III. The RI-R includes 22 items for self-report. It measures the frequency of post-traumatic symptoms in the previous four weeks. Subject are asked to note the frequency of symptoms on a scale from 0 (never) to 4 (most of the time). The measure of the severity of post-traumatic symptoms will be computed by summarizing 20 items on the questionnaire, as per Rodriguez et al (1999).

Functional impairment. This will be measured by means of items on the Diagnostic Predictive Scale (DPS), which relates to significant impairment in different areas of functioning (APA, 2000), for example: functioning in school, social relations, family relations, activity outside school and dangerous behavior. The participants will be asked to grade, on a scale of 0 (not at all) to 5 (very much) the degree to which they have experienced impairment in functioning in these areas. The severity of functioning impairment will be computed as the sum of all the items.

Exposure to traumatic events. This self-report questionnaire is a translation of the questionnaire by Ford et al. (1997), and works on the same basis. The subjects will be asked to answer, yes or no, whether they were ever exposed to one or more of 17 different traumatic events .

Strengths and difficulties. The Strength and Difficulties Questionnaire (SDQ), self-reported or filled out by parents, contains 25 items which assess different aspects of adjustment among children and adolescents focusing on behavioral symptoms. The questionnaire is intended to be completed by parents (or teachers) for children aged 3-16. Adolescents aged 11-16 can fill out the questionnaire by themselves (Goodman, 1997). The participants are asked to relate to 25 positive and negative statements, and respond as to what degree each statement fits their children, on a Likert scale of 1 (not true) to 3 (certainly true). The questionnaire is made up of five main factors: emotional symptoms, behavioral problems, attentiveness and hyperactivity, relations with the peer group, and pro-social behavior.

Children (Grades 3-6) Depression. Children Depression Inventory (CDI) (Kovacz, 1992) is a self-report questionnaire that assesses cognitive, affective, somatic and behavioral aspects of depression in children and adolescents from age 6 to 17. The original version of the questionnaire has 27 items, each containing three sentences. The child needs to choose the sentence that best describes his feelings over the previous two weeks. The scoring of the questionnaire presents a general score and five sub-scores: negative mood, interpersonal problems, ineffectiveness, anhedonia and self-image.

Anxiety. The Screen for Child Anxiety Related Emotional Disorders (SCARED), (Birmaher et al, 1997) is a self-report questionnaire that assesses anxiety symptoms in children. A general anxiety measure (eight items) and a separation anxiety measure (seven items) will be computed from the questionnaire. The subjects will be asked to grade, on a scale from 0 (generally not true) to 2 (generally true), the degree to which the items describes their situation. The general score on the two scales will be computed as the sum of the items.

Small children The report on the distress of small children in the family will be divided into two. For children aged 2-11, the parents will answer SDQs. For children aged 2-5, the parents will answer the Post-traumatic Stress Questionnaire. Each parent will answer a separate questionnaire.

Post-traumatic stress. The questionnaire is based on a semi-structured interview with the parents with respect to post-traumatic symptoms in their little children (ages 2-5) (Scheeringa & Zeanah, 1994). The parents will be asked to mark, on a scale of 0 (never) to 3 (yes), whether each one of the symptoms were evident in their children within the previous month.

ELIGIBILITY:
Inclusion Criteria:

* lost a son or daughter below the age of 18 as a result of a terrorist incident,
* at least six months previously

Exclusion Criteria:

* single-parent families
* family members who suffer from mental retardation, disturbances because of addiction, or psychiatric disturbance from the psychotic or autistic spectra (schizophrenia, manic-depressive illness, psychotic disturbances, PDD).

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Danny Brom, Ph.D, Study Director — The Israel Center for the Treatment of Psychotrauma
Locations (1):
- The Israel Center for the Treatment of Psychotrauma, Jerusalem, Israel